CLINICAL TRIAL: NCT04257721
Title: Development of a Predictive Score for Maxillary Osteochimionecrosis After Invasive Oral Surgery in Patients Treated Whith Biphosphonates or Biotherapies: the PREV-ONM Study
Brief Title: Predictive Score for Maxillary Osteonecrosis After Invasive Oral Surgery
Acronym: PREV-ONM
Status: Terminated | Type: Observational
Why Stopped: rate of inclusions too low
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01495-52
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Osteonecrosis Due to Drugs, Jaw
Keywords: jaw osteonecrosis; biphosphonates; antiangiogenic agents; oral surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Non-interventional prospective multicentre cohort study to determine a predictive score for the occurrence of osteochimionecrosis of the jaws after invasive oral surgery in patients who have received biphosphonates or antangiogenic drugs as part of chemotherapy with malignant bone disease (multiple myeloma or bone metastasis of a solid tumour).

Data are collected during the usual follow-up of patients during the first 3 months following surgery.

DETAILED DESCRIPTION:
Non-interventional prospective multicentre cohort study to determine a predictive score for the occurrence of osteochimionecrosis of the jaws after invasive oral surgery in patients who have received at least one of the following molecules as part of chemotherapy with malignant bone disease (multiple myeloma or bone metastasis of a solid tumour):

* Biphosphonates: ZOLEDRONATE (ZOMETA®), PAMIDRONATE (AREDIA®, OSTEPAM®)
* Anti-angiogenic: DENOSUMAB (XGEVA®), BEVACIZUMAB (AVASTIN®), RITUXIMAB (MABTHERA®, RIXATHON®, TRUXIMA®), SUNITINIB (SUTENT®), PAZOPANIB (VOTRIENT®), AXITINIB (INLYTA®), CARBOZANTINIB (CABOMETYX®, COMETRIQ®), SORAFENIB (NEXAVAR®)

The study protocol is based on the post-operative clinical and radiographic follow-up of patients. 3 consultations are scheduled:

* 1 week after surgery
* 1 month after surgery
* 3 months after surgery

The following information should be noted at each follow-up consultation:

* Appearance of gingival and mucosal tissues : normal or inflammatory physiological state
* Description of possible bone exposure: size, colour, spontaneous or induced bleeding
* Description and assessment of local pain
* Description of a local infection
* Results of a bacteriological sample in case of suppuration

The patient's participation in the study ends:

* at the end of one of the consultations at 1 week and 1 month as soon as osteochimionecrosis of the jaws is diagnosed by the investigating physician
* at the end of the consultation at 3 months otherwise
* in the event of the patient's death during the study
* in the event of the patient's renouncement to participate in the study The patient's participation period is therefore a maximum of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* patients who have received at least one of the following molecules as part of chemotherapy with malignant bone disease (multiple myeloma or bone metastasis of a solid tumour):
* Biphosphonates: ZOLEDRONATE (ZOMETA®), PAMIDRONATE (AREDIA®, OSTEPAM®)
* Anti-angiogenic: DENOSUMAB (XGEVA®), BEVACIZUMAB (AVASTIN®), RITUXIMAB (MABTHERA®, RIXATHON®, TRUXIMA®), SUNITINIB (SUTENT®), PAZOPANIB (VOTRIENT®), AXITINIB (INLYTA®), CARBOZANTINIB (CABOMETYX®, COMETRIQ®), SORAFENIB (NEXAVAR®)
* Patient who has had an oral surgical procedure (single or multiple dental extraction, with or without alveolectomy, under local or general anesthesia)

Exclusion Criteria:

* History of oral and/or cervico-facial radiotherapy
* Patient treated successively with biphosphonates and then with anti-angiogenic drugs.
* Patient under guardianship, curatorship, or imprisonment
* Patient who has notified his refusal to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have received biphosphonates or antangiogenic drugs as part of chemotherapy with malignant bone disease (multiple myeloma or bone metastasis of a solid tumour) and who has had an oral surgical procedure (single or multiple dental extraction, with or without alveolectomy, under local or general anesthesia)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
occurrence of osteonecrosis of the jaw | within 3 months after surgery
  occurrence of osteonecrosis of the jaw

SECONDARY OUTCOMES:
Frequency of post-operative healing (bone and gingival) and comparison to each patient's UCONNS score. | within 3 months after surgery
  Frequency of post-operative healing (bone and gingival) and comparison to each patient's UCONNS score.
  The UCONNS score was proposed in 2011. Its objective is to be able to predict the occurrence of osteochimionecrosis in conjunction with biphosphonate treatment before a dental invasive procedure (dental avulsions, implant placement, etc.). It takes into account several types of variables:
  * The patient's general condition and comorbidities (HIV, osteoporosis, rheumatoid arthritis, diabetes, presence or not of a soft tissue tumour, presence or not of a breast or prostate tumour, multiple myeloma, ...)
  * The nature, dose, and duration of use of the biphosphonate received
  * Oral hygiene
  * presence of suppuration, presence of osteomyelitis
  * The dental surgery received (endodontic treatment, periodontal treatment, surgery muco-gingival, tooth extraction, apical surgery, bone resection)

CONTACTS AND LOCATIONS:
Overall Officials: Emeline Noaillon, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (5):
- France (5):
  - Centre Hospitalier Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marx RE. Pamidronate (Aredia) and zoledronate (Zometa) induced avascular necrosis of the jaws: a growing epidemic. J Oral Maxillofac Surg. 2003 Sep;61(9):1115-7. doi: 10.1016/s0278-2391(03)00720-1. No abstract available. PMID 12966493
- [Background] Advisory Task Force on Bisphosphonate-Related Ostenonecrosis of the Jaws, American Association of Oral and Maxillofacial Surgeons. American Association of Oral and Maxillofacial Surgeons position paper on bisphosphonate-related osteonecrosis of the jaws. J Oral Maxillofac Surg. 2007 Mar;65(3):369-76. doi: 10.1016/j.joms.2006.11.003. No abstract available. PMID 17307580
- [Background] Ruggiero SL, Dodson TB, Fantasia J, Goodday R, Aghaloo T, Mehrotra B, O'Ryan F; American Association of Oral and Maxillofacial Surgeons. American Association of Oral and Maxillofacial Surgeons position paper on medication-related osteonecrosis of the jaw--2014 update. J Oral Maxillofac Surg. 2014 Oct;72(10):1938-56. doi: 10.1016/j.joms.2014.04.031. Epub 2014 May 5. PMID 25234529
- [Background] Qi WX, Tang LN, He AN, Yao Y, Shen Z. Risk of osteonecrosis of the jaw in cancer patients receiving denosumab: a meta-analysis of seven randomized controlled trials. Int J Clin Oncol. 2014 Apr;19(2):403-10. doi: 10.1007/s10147-013-0561-6. Epub 2013 Apr 20. PMID 23605142
- [Background] Allen MR, Burr DB. The pathogenesis of bisphosphonate-related osteonecrosis of the jaw: so many hypotheses, so few data. J Oral Maxillofac Surg. 2009 May;67(5 Suppl):61-70. doi: 10.1016/j.joms.2009.01.007. PMID 19371816
- [Background] Gaudin E, Seidel L, Bacevic M, Rompen E, Lambert F. Occurrence and risk indicators of medication-related osteonecrosis of the jaw after dental extraction: a systematic review and meta-analysis. J Clin Periodontol. 2015 Oct;42(10):922-32. doi: 10.1111/jcpe.12455. Epub 2015 Nov 3. PMID 26362756
- [Background] Peddi P, Lopez-Olivo MA, Pratt GF, Suarez-Almazor ME. Denosumab in patients with cancer and skeletal metastases: a systematic review and meta-analysis. Cancer Treat Rev. 2013 Feb;39(1):97-104. doi: 10.1016/j.ctrv.2012.07.002. Epub 2012 Aug 13. PMID 22898302
- [Background] Landesberg R, Woo V, Cremers S, Cozin M, Marolt D, Vunjak-Novakovic G, Kousteni S, Raghavan S. Potential pathophysiological mechanisms in osteonecrosis of the jaw. Ann N Y Acad Sci. 2011 Feb;1218:62-79. doi: 10.1111/j.1749-6632.2010.05835.x. PMID 21291478
- [Background] Reich W, Bilkenroth U, Schubert J, Wickenhauser C, Eckert AW. Surgical treatment of bisphosphonate-associated osteonecrosis: Prognostic score and long-term results. J Craniomaxillofac Surg. 2015 Nov;43(9):1809-22. doi: 10.1016/j.jcms.2015.07.035. Epub 2015 Aug 6. PMID 26321065